CLINICAL TRIAL: NCT06365554
Title: Safety and Feasibility of On-Premise and Remote Robotic Neurointervention
Brief Title: On-Premise and Remote Robotic Neurointervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Remedy Robotics, Inc. (Industry)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Cerebrovascular Disease
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Group undergoing intervention with the Remedy Robot.
  Interventions: Device: Remedy Robot

INTERVENTIONS:
Device: Remedy Robot — A trained Neurointerventionalist will operate the Remedy Robot from a computer-based user interface in a room adjacent to the patient. An entire cerebral angiogram or cerebral embolization will be performed, excluding insertion and removal of the femoral sheath.

SUMMARY:
This study is a prospective, single arm, single-center study to evaluate the safety and feasibility of the Remedy Robot for on premise and remote robotic Neurointervention.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-center study to evaluate the safety and effectiveness of the Remedy Robot for patients with a clinical indication for Neurointervention.

ELIGIBILITY:
Inclusion criteria

* The patient is ≥ 18 years of age
* The Investigator deems the patient appropriate for manual and robotic-assisted Neurointervention.
* The patient or their substitute decision-maker has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent.

Exclusion criteria:

* Patients currently pregnant or breastfeeding.
* People with any of the following vascular history:
* Known congenital aortopathy, connective tissue disorder or vasculopathy
* Known arterial dissection of any kind
* Bleeding diathesis
* Use of Warfarin, IV Heparin, Clexane, Fondaparinux or any new oral anticoagulants (NOACs) or direct oral anticoagulants (DOACs)

People with any of the following medical history:

* Active malignancy
* Known contrast allergy
* Height > 190cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Procedural safety | Measured from the start of the procedure through 24 hours or discharge
  Incidence of intra- and peri-procedural events, including all cause mortality, stroke, arterial dissection, arterial perforation
Procedural Technical Success | Measured from the start of the procedure through to the completion of the procedure
  Successful completion of the robotic-assisted endovascular procedure absent any unplanned conversion to manual control

IPD SHARING:
Plan to Share IPD: No